CLINICAL TRIAL: NCT05181111
Title: Continuous Monitoring of Patients in and After the Acute Admission Ward to Optimize Clinical Pathways
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rijnstate Hospital (Other)
Collaborators: University of Twente (Other); Philips Research Eindhoven (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LHC 2021-1838
Record Dates: First submitted 2021-12-23; First posted 2022-01-06 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Monitoring; Clinical Deterioration; Acute Disease
Keywords: prediction; acute admission ward; continuous monitoring
MeSH Terms: conditions — Clinical Deterioration; Acute Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monitoring Group (Experimental): wearable sensor, besides usual care monitoring
  Interventions: Device: Wearable Sensor; Other: Usual Care
- Usual Care group (Other): usual care monitoring
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: Wearable Sensor — The sensor measures vital signs including heart rate and respiratory rate, posture and level of physical activity.
  Other Names: Philips Healthdot
  Arms: Monitoring Group
Other: Usual Care — Usual Care Monitoring

SUMMARY:
Hospitals aim to hospitalize patients when necessary and discharge patients when possible. However, the triage process and discharge management of patients in e.g. the Acute Admission Ward, is not a trivial task. The upcoming technology of wearable monitoring devices, whereby patients can be continuously monitored with an unobtrusive vital signs device, might help getting more insight into patients' health condition and thus help facilitate efficient and effective triaging.

Therefore, the primary objective is to assess the effects of continuous monitoring of patients in the acute admission ward (AAW) on the percentage of patients who can be discharged home. Secondary objectives are to assess the length of stay in the acute admission ward and in the in-hospital wards, as well as the effect on admission to the intensive care unit, rapid response team calls and hospital readmission. The predictive value of algorithms applied to the monitoring data combined with other parameters to detect timely deterioration and predict discharge will be assessed. Facilitators and barriers for implementing such a system will be investigated.

ELIGIBILITY:
Inclusion Criteria:

In order for a patient to be eligible to participate in this study, the following criteria need to be met:

* admitted to the AAW
* Age ≥ 18 years
* Able to speak and read Dutch
* Willing and able to provide written informed consent

Exclusion Criteria:

A patient who meets any of the following criteria will be excluded from participation:

* Not able or willing to wear a wearable sensor on the chest continuously for 14 days
* Planned major surgery in the upcoming 30 days
* At the time of AAW admission already known to be discharged home or admitted to the hospital
* Any skin condition, for example prior rash, discoloration, scars, infection, injury or open wounds at the area (Left lower rib) where the sensor needs to be placed
* Known sensitivity to medical adhesives
* Wearing an active implantable device (e.g. ICD, pacemaker)
* Intend to go to the sauna or go swimming in the upcoming 14 days
* Pregnant or breastfeeding
* Use of creams or lotions that are known to influence the skin at the area where sensor is placed (such as medical and non-medical creams or lotions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-12-05 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients discharged home from acute admission ward | up to 7 days
  Percentage of patients discharged home from acute admission ward

SECONDARY OUTCOMES:
Length of stay in the acute admission ward | up to 7 days
  Length of stay in the acute admission ward
Length of stay in the in-hospital wards | up to 31 days
  Length of stay in the in-hospital wards
Percentage of Rapid Response Team calls | up to 31 days
  Percentage of Rapid Response Team calls
Percentage of Intensive Care Unit Admissions | up to 31 days
  Percentage of Intensive Care Unit Admissions
Percentage of unplanned readmissions to the hospitals | up to 31 days
  Percentage of unplanned readmissions to the hospitals

OTHER OUTCOMES:
Deterioration | up to 7 days
  Deterioration will be assessed using clinical data
Facilitators and Barriers for implementing continuous monitoring system (interviews) | up to 31 days
  Facilitators and Barriers for implementing continuous monitoring system in practice (interviews with stakeholders)

CONTACTS AND LOCATIONS:
Overall Officials: Carine JM Doggen, Prof PhD, Principal Investigator — Rijnstate Hospital
Locations (1):
- Rijnstate Hospital, Arnhem, Netherlands

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Kant N, Garssen SH, Vernooij CA, Mauritz GJ, Koning MV, Bosch FH, Doggen CJM. Enhancing discharge decision-making through continuous monitoring in an acute admission ward: a randomized controlled trial. Intern Emerg Med. 2024 Jun;19(4):1051-1061. doi: 10.1007/s11739-024-03582-y. Epub 2024 Apr 15. PMID 38619713
- [Derived] Garssen SH, Kant N, Vernooij CA, Mauritz GJ, Koning MV, Bosch FH, Doggen CJM. Continuous monitoring of patients in and after the acute admission ward to improve clinical pathways: study protocol for a randomized controlled trial (Optimal-AAW). Trials. 2023 Jun 15;24(1):405. doi: 10.1186/s13063-023-07416-8. PMID 37316919